CLINICAL TRIAL: NCT07370545
Title: The Influence of Shade Guide Presentation Sequence and Psychosocial Factors on Patient Tooth Shade Selection: A Three-Arm Randomized Controlled Trial
Brief Title: Impact of Presentation Sequence on Patient Tooth Shade Selection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alaa Al-Haddad, Clinical Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2/5/1/175
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Shade Match; Teeth Color; Patient Preference; Aesthetic Perception
Keywords: Patient Preference; shade guide; teeth color; shade selection
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Sequential Presentation (Natural then Bleached) (Experimental): Participants in this arm will undergo a two-phase shade selection process. In Phase 1, they will select their preferred tooth shade from the natural range of the VITA 3D-Master shade guide (1M1 to 5M3). In Phase 2, the bleached shade tabs (0M1 to 0M3) will be introduced, and participants will be asked if they wish to maintain or alter their initial selection. The final choice and the magnitude of change (Delta L*) will be recorded.
  Interventions: Behavioral: Sequential Shade Presentation (Natural to Bleached)
- Group B: Sequential Presentation (Bleached then Natural) (Experimental): Participants in this arm will undergo a two-phase shade selection process. In Phase 1, they will select their preferred tooth shade from the bleached range of the VITA 3D-Master shade guide (0M1 to 0M3). In Phase 2, the full natural range (1M1 to 5M3) will be introduced, and participants will be asked if they wish to maintain or alter their initial selection. This arm serves to measure the "order effect" in the opposite direction of Group A.
  Interventions: Behavioral: Sequential Shade Presentation (Bleached to Natural)
- Group C: Simultaneous Presentation (Full Range) (Active Comparator): Participants in this arm will undergo a single-phase shade selection process. They will be presented with the full range of the VITA 3D-Master shade guide, including both natural (1M1 to 5M3) and bleached (0M1 to 0M3) tabs, simultaneously. This arm serves as the control baseline to determine patient preference in the absence of sequential presentation bias.
  Interventions: Behavioral: Simultaneous Shade Presentation (Full Range)

INTERVENTIONS:
Behavioral: Sequential Shade Presentation (Natural to Bleached) — Participants are first presented with the natural range of the VITA 3D-Master shade guide (1M1-5M3) to select an initial preference. Following this, the bleached shade tabs (0M1-0M3) are introduced, and participants are invited to finalize their choice. This procedure measures the "pull" toward lighter shades when introduced as a secondary option.
  Arms: Group A: Sequential Presentation (Natural then Bleached)
Behavioral: Sequential Shade Presentation (Bleached to Natural) — Participants are first presented with the bleached range of the VITA 3D-Master shade guide (0M1-0M3) to select an initial preference. Following this, the full natural range (1M1-5M3) is introduced, and participants are invited to finalize their choice. This procedure measures the stability of the bleached shade preference when natural alternatives are subsequently provided.
  Arms: Group B: Sequential Presentation (Bleached then Natural)
Behavioral: Simultaneous Shade Presentation (Full Range) — Participants are presented with the complete VITA 3D-Master shade guide, including both natural (1M1-5M3) and bleached (0M1-0M3) tabs, in a single session. Participants select their preferred shade from the entire range simultaneously. This serves as the control method to establish baseline preference without sequential bias.
  Arms: Group C: Simultaneous Presentation (Full Range)

SUMMARY:
This study is a clinical trial designed to understand how the way a dentist presents tooth color options affects a patient's final choice for their dental treatment. The insvestigators know that patients often prefer lighter, "bleached" shades, but the process of choosing can be influenced by the order in which the shades are shown.

The insvestigators will randomly dividing participants into three groups. One group will see natural shades first, followed by bleached shades. A second group will see bleached shades first, followed by natural shades. The third group will see all shades at once.

The main goal is to measure how often patients change their mind (switch their choice) and by how much (the "jump" in lightness) depending on the order of presentation. The insvestigators will also use a questionnaire to see if a patient's self-consciousness about their smile affects how light of a shade they choose. The results will help dentists improve communication and ensure patients are truly satisfied with their final aesthetic decision.

DETAILED DESCRIPTION:
This is a prospective, single-center, three-arm parallel-group Randomized Controlled Trial (RCT) designed to rigorously investigate the cognitive bias known as the "order effect" in patient-driven tooth shade selection. The study aims to quantify the influence of sequential versus simultaneous shade guide presentation on final aesthetic preference and to correlate this choice with the patient's underlying psychosocial perception of their dental aesthetics.

Methodology: Participants seeking aesthetic dental treatment will be randomized (1:1:1) into three intervention groups:

1. Group A (Natural -> Bleached): Sequential presentation of natural shades followed by the introduction of bleached shades.
2. Group B (Bleached -> Natural): Sequential presentation of bleached shades followed by the introduction of natural shades.
3. Group C (Simultaneous): Single presentation of the full VITA 3D-Master shade guide (natural and bleached tabs combined).

Outcome Measures: The primary outcomes are the switching frequency and the magnitude of change (Delta L*) between initial and final selections in the sequential groups (A and B), and the comparison of the final proportion of bleached shade selections across all three groups. Secondary outcomes include the correlation between the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ) total score and the final selected shade's L* value, and the quantification of the Patient-Clinician Discrepancy using CIE Delta E00 between the patient's choice and an independent clinician's recommendation.

Significance: This study will provide evidence-based guidelines for clinical practice, moving beyond anecdotal preference recording to a structured, bias-mitigating approach to shared aesthetic decision-making. The integration of the PIDAQ and objective colorimetric analysis (Lab*) and Delta E00 will provide a novel, high-impact explanation for the observed preference for lighter shades.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Seeking aesthetic dental treatment (e.g., anterior restorations, veneers, or tooth bleaching).
* Possessing at least one sound, non-restored maxillary central incisor (tooth #8 or #9) to serve as a reference for objective shade measurement.
* Ability to understand the study procedures and provide written informed consent.
* Fluent in the language of the study (Arabic/English) to complete the psychosocial questionnaire (PIDAQ).

Exclusion Criteria:

* Congenital or acquired color vision deficiencies (screened using the Ishihara test).
* Cognitive impairments or psychological conditions that may affect decision-making or the ability to complete questionnaires.
* Extensive existing restorations, crowns, or severe intrinsic staining (e.g., tetracycline staining) on the maxillary anterior teeth.
* Active periodontal disease or poor oral hygiene that may interfere with accurate shade assessment.
* Previous history of professional tooth bleaching within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Final Shade Selection (L* Value) | At the time of shade selection (Day 1)
  The lightness (L*) value of the final tooth shade selected by the patient using the VITA 3D-Master guide. The VITA 3D-Master tabs will be converted to CIE Lab* coordinates based on established conversion tables. This measure assesses the final aesthetic preference across the three randomized groups.
Switching Frequency | At the time of shade selection (Day 1)
  The percentage of participants in the sequential groups (Group A and Group B) who change their initial shade selection after the second range of shade tabs is introduced. This measures the stability of the initial choice and the susceptibility to presentation bias.

SECONDARY OUTCOMES:
Magnitude of Shade Change (Delta L*) | At the time of shade selection (Day 1)
  The numerical difference in lightness (L*) between the patient's initial shade selection and their final shade selection in the sequential groups (Group A and Group B). A positive value indicates a "jump" toward a lighter shade, while a negative value indicates a shift toward a darker shade.
Psychosocial Impact Correlation (PIDAQ) | Baseline (Day 1)
  The correlation coefficient between the total score of the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ) and the final selected shade's L* value. Higher PIDAQ scores indicate a greater negative psychosocial impact of dental aesthetics.
Patient-Clinician Discrepancy (Delta E00) | At the time of shade selection (Day 1)
  The color difference (calculated using the CIE Delta E00 formula) between the patient's final selected shade tab and the independent clinician's professional recommendation. This quantifies the gap between patient desire and professional aesthetic judgment.
Objective Color Discrepancy (Delta E00) | At the time of shade selection (Day 1)
  The color difference (calculated using the CIE Delta E 00 formula) between the patient's final selected shade tab and the objective natural tooth color measured by a spectrophotometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Jordan Hospital, Dental Department, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
annonmous shade selected by participant and clinican, with PIDAQ total scores.
Supporting Information: Study Protocol, SAP, ICF, CSR